CLINICAL TRIAL: NCT02053493
Title: Nitrate's Effect on Activity Tolerance in Heart Failure With Preserved Ejection Fraction
Acronym: NEAT-HFpeF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adrian Hernandez (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Mayo Clinic (Other); University of Vermont (Other)
Responsible Party: Sponsor-Investigator, Adrian Hernandez, Professor of Medicine, DUMC; Director, Health Services and Outcomes Research, DCRI, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00050042; 4U10HL084904-10 (NIH)
Record Dates: First submitted 2014-01-03; First posted 2014-02-03 (Estimated); Results first posted 2016-11-28 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure
Keywords: Heart Failure; Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isosorbide Mononitrate (Active Comparator): Isosorbide Mononitrate with dose up-titration (30 to 120 mg/day over 4 weeks)
  Interventions: Drug: Isosorbide Mononitrate
- Isosorbide Mononitate Placebo (Placebo Comparator): Isosorbide Mononitrate placebo with dose up-titration (30 to 120 mg/day over 4 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isosorbide Mononitrate — Dispense phase 1 study drug:
  Weeks 1 and 2: No study drug (baseline) Week 3: 30 mg ISMN Week 4: 60 mg ISMN Weeks 5 and 6: 120 mg ISMN
  Dispense phase-2 study drug:
  Weeks 7 and 8: No study drug (washout) Week 9: 30 mg ISMN Week 10: 60 mg ISMN Weeks 11 and 12: 120 mg ISMN
  Other Names: Imdur, ISMO, Monoket
  Arms: Isosorbide Mononitrate
Drug: Placebo — Dispense phase 1 study drug:
  Weeks 1 and 2: No study drug (baseline) Week 3: 30 mg Placebo Week 4: 60 mg Placebo Weeks 5 and 6: 120 mg Placebo
  Dispense phase-2 study drug:
  Weeks 7 and 8: No study drug (washout) Week 9: 30 mg Placebo Week 10: 60 mg Placebo Weeks 11 and 12: 120 mg Placebo
  Arms: Isosorbide Mononitate Placebo

SUMMARY:
A randomized, double-blinded, placebo-controlled crossover study to assess effect of isosorbide mononitrate with dose up-titration on activity tolerance as assessed by (hip-worn, tri-axial) accelerometry.

DETAILED DESCRIPTION:
To evaluate whether isosorbide mononitrate increases daily activity as assessed by 14-day averaged arbitrary accelerometry units in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years
2. Symptoms of dyspnea (NYHA class II-IV) without evidence of a non-cardiac or ischemic explanation for dyspnea
3. Ejection fraction (EF) ≥ 50% as determined on imaging study within 12 months of enrollment with no change in clinical status suggesting potential for deterioration in systolic function
4. Stable medical therapy for 30 days as defined by:

   * No addition or removal of ACE, Angiotensin receptor blockers (ARBs), beta-blockers, calcium channel blockers (CCBs) or aldosterone antagonists
   * No change in dosage of ACE, ARBs, beta-blockers,CCBs or aldosterone antagonists of more than 100%
5. One of the following within the last 12 months

   * Previous hospitalization for heart failure (HF) with radiographic evidence of pulmonary congestion (pulmonary venous hypertension, vascular congestion, interstitial edema, pleural effusion) or
   * Catheterization documented elevated filling pressures at rest (LVEDP≥15 or PCWP≥20) or with exercise (PCWP≥25) or
   * Elevated NT-proBNP (> 400 pg/ml) or BNP (> 200 pg/ml) or
   * Echo evidence of diastolic dysfunction / elevated filling pressures (at least two) E/A > 1.5 + decrease in E/A of > 0.5 with valsalva Deceleration time ≤ 140 ms Pulmonary vein velocity in systole < diastole (PVs<PVd)sinus rhythm) E/e'≥15 Left atrial enlargement (≥ moderate) Pulmonary artery systolic pressure > 40 mmHg Evidence of left ventricular hypertrophy
   * LV mass/BSA ≥ 96 (♀) or ≥ 116 (♂) g/m2
   * Relative wall thickness ≥ 0.43 (♂ or ♀) [(IVS+PW)/LVEDD]
   * Posterior wall thickness ≥ 0.9 (♀) or 1.0 (♂) cm
6. No chronic nitrate therapy or infrequent (≤ 1x week) use of intermittent sublingual nitroglycerin within last 3 months
7. Ambulatory (not wheelchair / scooter / walker / cane dependent)
8. HF is the primary factor limiting activity as indicated by answering # 2 to the following question:

My ability to be active is most limited by:

1. Joint, foot, leg, hip or back pain
2. Shortness of breath and/or fatigue and/or chest pain
3. Unsteadiness or dizziness
4. Lifestyle, weather, or I just don't like to be active

9. Body size allows wearing of the accelerometer belt as confirmed by ability to comfortably fasten the test belt provided for the screening process (belt designed to fit persons with BMI 20-40 Kg/m2 but belt may fit some persons outside this range)

10. Willingness to wear the accelerometer belt for the duration of the trial 11. Willingness to provide informed consent

Exclusion Criteria:

1. Recent (< 3 months) hospitalization for HF
2. Hemoglobin < 8.0 g/dl
3. Glomerular filtration rate < 20 ml/min/1.73 m2 on most recent clinical laboratories
4. SBP < 110 mmHg or > 180 mmHg at consent
5. Diastolic blood pressure < 40 mmHg or > 100 mmHg at consent
6. Resting HR > 110 bpm at consent
7. Previous adverse reaction to nitrates necessitating withdrawal of therapy
8. Chronic therapy with phosphodiesterase type-5 inhibitors (intermittent use of phosphodiesterase type-5 inhibitors for erectile dysfunction is allowable if the patient is willing to hold for the duration of the trial)
9. Regularly (> 1x per week) swims or does water aerobics
10. Significant COPD thought to contribute to dyspnea
11. Ischemia thought to contribute to dyspnea
12. Documentation of previous EF < 50%
13. Acute coronary syndrome within 3 months defined by electrocardiographic changes and biomarkers of myocardial necrosis (e.g. troponin) in an appropriate clinical setting (chest discomfort or anginal equivalent)
14. Percutaneous coronary intervention, coronary artery bypass grafting or new biventricular pacing within past 3 months
15. Primary hypertrophic cardiomyopathy
16. Infiltrative cardiomyopathy (amyloid)
17. Constrictive pericarditis or tamponade
18. Active myocarditis
19. Complex congenital heart disease
20. Active collagen vascular disease
21. More than mild aortic or mitral stenosis
22. Intrinsic (prolapse, rheumatic) valve disease with moderate to severe or severe mitral, tricuspid or aortic regurgitation
23. Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment
24. Terminal illness (other than HF) with expected survival of less than 1 year
25. Enrollment or planned enrollment in another therapeutic clinical trial in the next 3 months
26. Inability to comply with planned study procedures
27. Pregnant women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Anstrom, PhD, Principal Investigator — Duke Clinical Research Institute; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (22):
- United States (22):
  - Christiana Care Health Services, Newark, Delaware
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston V.A. Healthcare System, West Roxbury, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Metro Health System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Michael E Debakey VA Medical Center, Houston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah
  - V.A. Medical Center, Salt Lake City, Utah
  - The University of Vermont - Fletcher Allen Health Care, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
After the study results have been published, site-specific participant data will be shared with sites upon request. Sites are expected to follow their specific institutional policies regarding sharing results with their participants.

REFERENCES:
- [Derived] Reddy YNV, Rikhi A, Obokata M, Shah SJ, Lewis GD, AbouEzzedine OF, Dunlay S, McNulty S, Chakraborty H, Stevenson LW, Redfield MM, Borlaug BA. Quality of life in heart failure with preserved ejection fraction: importance of obesity, functional capacity, and physical inactivity. Eur J Heart Fail. 2020 Jun;22(6):1009-1018. doi: 10.1002/ejhf.1788. Epub 2020 Mar 9. PMID 32150314
- [Derived] Snipelisky D, Kelly J, Levine JA, Koepp GA, Anstrom KJ, McNulty SE, Zakeri R, Felker GM, Hernandez AF, Braunwald E, Redfield MM. Accelerometer-Measured Daily Activity in Heart Failure With Preserved Ejection Fraction: Clinical Correlates and Association With Standard Heart Failure Severity Indices. Circ Heart Fail. 2017 Jun;10(6):e003878. doi: 10.1161/CIRCHEARTFAILURE.117.003878. PMID 28588021
- [Derived] Redfield MM, Anstrom KJ, Levine JA, Koepp GA, Borlaug BA, Chen HH, LeWinter MM, Joseph SM, Shah SJ, Semigran MJ, Felker GM, Cole RT, Reeves GR, Tedford RJ, Tang WH, McNulty SE, Velazquez EJ, Shah MR, Braunwald E; NHLBI Heart Failure Clinical Research Network. Isosorbide Mononitrate in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2015 Dec 10;373(24):2314-24. doi: 10.1056/NEJMoa1510774. Epub 2015 Nov 8. PMID 26549714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients admitted to the participating HFN centers with signs and symptoms suggestive of HFpEF will be screened including their ability to wear the accelerometer belt. Patients meeting eligibility criteria will be approached regarding participation in this study.
Pre-assignment Details: All subjects who fulfill all the inclusion criteria and none of the exclusion criteria will undergo the baseline studies and then be randomized.
Groups:
- Isosorbide Mononitrate Crossover to Placebo: Isosorbide Mononitrate with dose up-titration (30 to 120 mg/day over 4 weeks)
  Isosorbide Mononitrate: Dispense phase 1 study drug:
  Weeks 1 and 2: No study drug (baseline) Week 3: 30 mg ISMN Week 4: 60 mg ISMN Weeks 5 and 6: 120 mg ISMN
  Dispense phase-2 study drug:
  Weeks 7 and 8: No study drug (washout) Week 9: 30 mg ISMN Week 10: 60 mg ISMN Weeks 11 and 12: 120 mg ISMN
- Placebo Crossover to Isosorbide Mononitrate: Isosorbide Mononitrate placebo with dose up-titration (30 to 120 mg/day over 4 weeks)
  Placebo: Dispense phase 1 study drug:
  Weeks 1 and 2: No study drug (baseline) Week 3: 30 mg Placebo Week 4: 60 mg Placebo Weeks 5 and 6: 120 mg Placebo
  Dispense phase-2 study drug:
  Weeks 7 and 8: No study drug (washout) Week 9: 30 mg Placebo Week 10: 60 mg Placebo Weeks 11 and 12: 120 mg Placebo
Period: Overall Study
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Started | 51 | 59
Completed | 50 | 58
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate | Total
Number analyzed (Participants) | 51 | 59 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (8.7) | 68.8 (9.7) | 69.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 38 | 63
  Male | 26 | 21 | 47
Region of Enrollment [Number; unit: participants]
  United States | 51 | 59 | 110

OUTCOME MEASURES:

1. Primary Outcome: Arbitrary Accelerometry Units (AAU) (Phase I)
Description: To evaluate whether isosorbide mononitrate increases daily activity as assessed by 14-day averaged arbitrary accelerometry units in comparison to placebo. An arbitrary accelerometer unit is calculated within the accelerometer device that is worn by the patient and represents level of activity based on patient movement. Higher values indicate more movement. 0 indicates no movement.
Time Frame: 5-6 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 45 | 56
accelerometry units | 9370 (4601) | 9538 (6286)

2. Secondary Outcome: Six Minute Walk Distance (Phase I)
Description: To evaluate whether isosorbide mononitrate (ISMN) improves functional capacity by 6 minute walk distance in comparison to placebo.
Time Frame: Week 7
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 49 | 57
meters | 307.8 (125.5) | 327.1 (126.0)

3. Secondary Outcome: Six Minute Walk Distance (Phase II)
Description: as for outcome 2
Time Frame: Week 13
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 47 | 57
meters | 321.3 (132.4) | 329.7 (132.1)

4. Secondary Outcome: Patient Preference for Isosorbide Mononitrate Treatment at the End of Study.
Description: Self reported participant preference for study period 1 vs. study period 2.
Time Frame: Week 13
Population: Participants with usable data included in the results
Measure: Number; unit: participants
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 48 | 57
participants
  Phase1 | 14 | 14
  Phase2 | 18 | 24
  No Preference | 16 | 19

5. Secondary Outcome: Borg Score During 6 Minute Walk Test (Phase I)
Description: To evaluate whether isosorbide mononitrate improves quality of life in comparison to placebo. The Borg Scale consists of scale range of 0 to 10 (where 0 indicates no breathlessness at all and 10 indicates maximum breathlessness). Lower values are considered to be better than higher values.
Time Frame: Week 7
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 44 | 52
units on a scale | 4.1 (2.6) | 4.0 (2.2)

6. Secondary Outcome: Borg Score During 6 Minute Walk Test (Phase II)
Description: as for outcome 5
Time Frame: Week 13
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 40 | 49
units on a scale | 3.8 (2.3) | 3.8 (2.0)

7. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire Overall Summary Score (Phase I)
Description: To evaluate whether isosorbide mononitrate improves quality of life in comparison to placebo. The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, fewer symptoms, better quality of life).
Time Frame: Week 7
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 50 | 58
units on a scale | 57.3 (23.4) | 64.2 (24.2)

8. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire Overall Summary Score (Phase II)
Description: To evaluate whether isosorbide mononitrate improves quality of life in comparison to placebo. • The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (eg, better functioning, fewer symptoms, better quality of life).Higher values of the overall KCCQ score are considered to be better than lower values.
Time Frame: Week 13
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 49 | 58
units on a scale | 59.1 (23.6) | 61.6 (23.5)

9. Primary Outcome: Arbitrary Accelerometry Units (AAU) (Phase II)
Description: as for outcome 1
Time Frame: 11-12 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 42 | 49
accelerometry units | 8824 (3877) | 8900 (5457)

10. Secondary Outcome: N-terminal Pro-B-type Natriuretic Peptide Level (Phase I)
Description: To evaluate whether isosorbide mononitrate improves natriuretic peptide levels in comparison to placebo
Time Frame: Week 7
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 49 | 57
pg/mL | 513.0 (803.2) | 542.4 (710.9)

11. Secondary Outcome: N-terminal Pro-B-type Natriuretic Peptide Level (Phase II)
Description: To evaluate whether isosorbide mononitrate improves natriuretic peptide levels in comparison to placebo
Time Frame: Week 13
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 47 | 54
pg/mL | 466.1 (677.4) | 573.3 (756.1)

12. Secondary Outcome: Improvement in Daily Activity - Hours Active Per Day (Phase I)
Description: To evaluate whether isosorbide mononitrate in comparison to placebo improves daily activity as measured by Hours active per day during maximal dose of study drug
Time Frame: 5-6 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 45 | 56
Hours/day | 9.4 (2.4) | 9.1 (2.4)

13. Secondary Outcome: Improvement in Daily Activity - Hours Active Per Day (Phase II)
Description: as for outcome 12
Time Frame: 11-12 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: Hours/day
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 42 | 49
Hours/day | 9.4 (2.4) | 8.8 (2.5)

14. Secondary Outcome: Improvement in Daily Activity - Slope of Daily Average (Phase I)
Description: To evaluate whether isosorbide mononitrate in comparison to placebo improves daily activity as measured by Slope of daily averaged arbitrary accelerometry units during study drug administration. An arbitrary accelerometer unit is calculated within the accelerometer device that is worn by the patient and represents level of activity based on patient movement. Higher values indicate more movement. 0 indicates no movement.
Time Frame: 3-6 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units/day
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 47 | 58
accelerometry units/day | -3.4 (23.1) | -1.3 (26.9)

15. Secondary Outcome: Improvement in Daily Activity - Slope of Daily Average (Phase II)
Description: as for outcome 14
Time Frame: 9-12 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units/day
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 42 | 53
accelerometry units/day | 2.6 (20.1) | -3.9 (16.4)

16. Secondary Outcome: Improvement in Daily Activity - Area Under the Curve (Phase I)
Description: To evaluate whether isosorbide mononitrate in comparison to placebo improves daily activity as measured by Area under the curve (AUC) of arbitrary accelerometry units during study drug administration. An arbitrary accelerometer unit is calculated within the accelerometer device that is worn by the patient and represents level of activity based on patient movement. Higher values indicate more movement. 0 indicates no movement. Area under the curve is defined as ((7*average acceleromtery units/day during 30 mg) + (7*average acceleromtery units/day during 60 mg) + (14*average acceleromtery units/day during 120 mg))/28
Time Frame: 3-6 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 39 | 54
accelerometry units | 9621.4 (4367.8) | 9714.0 (6273.6)

17. Secondary Outcome: Improvement in Daily Activity - Area Under the Curve (Phase II)
Description: as for outcome 16
Time Frame: 9-12 weeks
Population: Participants with usable data included in the results
Measure: Mean (Standard Deviation); unit: accelerometry units
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Number analyzed (Participants) | 38 | 44
accelerometry units | 9146.5 (3695.3) | 9325.9 (5668.2)

ADVERSE EVENTS:
Time Frame: Informed Consent through Week 15 phone visit
Description: Per protocol, non-serious AEs were not collected; all SAEs were collected except for anticipated, disease-related events in patients with HF with preserved EF.
  3 time points summarized: Informed Consent to start of Phase 1 study drug, Phase 1 study drug start to start of Phase 2 study drug, Phase 2 study drug start to Week 15 phone call.
Arm/Group | Isosorbide Mononitrate Crossover to Placebo | Placebo Crossover to Isosorbide Mononitrate
Serious Adverse Events (participants affected / at risk) | 2/51 | 1/59
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isosorbide Mononitrate Crossover to Placebo (N=51) | Placebo Crossover to Isosorbide Mononitrate (N=59)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Phase 1 study drug start to start of Phase 2 study drug
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Phase 2 study drug start to Week 15 phone call
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) — Phase 2 study drug start to Week 15 phone call
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) — Informed consent to start of phase 1 study drug
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) — Informed consent to start of phase 1 study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less